CLINICAL TRIAL: NCT05743647
Title: Assessment of Brain Activation With Different Mirror Therapy Tasks - Contribution of EEG and fNIRS in Healthy Subjects.
Brief Title: Study of Cerebral Activation During Different Rehabilitation Tasks of Lower Limb in Virtual Mirror Therapy in Healthy Subjects
Acronym: ARTHEMIRS2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2022-06
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Virtual Mirror therapy; Electroencephalography; Near infrared spectroscopy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young: 40 right handed healthy subject aged between 18 and 40
  Interventions: Device: Observation (OBS); Device: Observation and imagination (OBS-IM); Device: Observation and realization (OBS-REAL)
- Old: 40 right handed healthy subject aged between 41 and 75
  Interventions: Device: Observation (OBS); Device: Observation and imagination (OBS-IM); Device: Observation and realization (OBS-REAL)

INTERVENTIONS:
Device: Observation (OBS) — Subject is seated in a chair facing IVS4. He places his right lower under the screen. The flexion / extension movement of the ankle at a frequency of 0.5 Hz is then recorded. Then for the "mirror" effect the software reverses the recorded movement, the lower right limb becomes the lower left limb on the screen.
  The subject only observe the movement on the screen during the recordings. The subject does not produce any movement.
Device: Observation and imagination (OBS-IM) — Subject is seated in a chair facing IVS4. He places his right lower under the screen. The flexion / extension movement of the ankle at a frequency of 0.5 Hz is then recorded. Then for the "mirror" effect the software reverses the recorded movement, the lower right limb becomes the lower left limb on the screen.
  The subject observe the movement but also imagine to realized it.
Device: Observation and realization (OBS-REAL) — Subject is seated in a chair facing IVS4. He places his right lower under the screen. The flexion / extension movement of the ankle at a frequency of 0.5 Hz is then recorded. Then for the "mirror" effect the software reverses the recorded movement, the lower right limb becomes the lower left limb on the screen.
  The subject observe the movement on the screen and realized it

SUMMARY:
The purpose of this study is to investigate the cerebral activation during visual motor simulation in healthy subjects in 3 conditions: observation (OBS), observation and imagination (OBS-IM) and observation and realization (OBS-REAL). The investigators goal is to compare cerebral activation during the three different tasks using EEG and fNIRS.

DETAILED DESCRIPTION:
Mirror therapy is a rehabilitation technique that has been shown to be effective in restoring upper limb motor skills in patients with stroke. However, it comes up against certain constraints of clinical use such as installation difficulties or the obligation of symmetrical bilateral work. These constraints can be limited by the use of so-called 2nd generation virtual mirror therapy technologies. It is therefore likely that these new technologies will improve the feasibility and effectiveness of mirror therapy in rehabilitation.

The brain mechanisms involved in virtual mirror therapy are not yet fully understood. EEG (Electroencephalography) and fNIRS (functional Near Infra Red Spectroscopy) are two functional method that allows to study the cerebral cortex changes during different tasks (like fMRI).

These techniques therefore makes it possible to study brain activation under more ecological conditions than fMRI and are therefore particularly suitable for exploring rehabilitation techniques.

This research aims to study and compare in healthy subjects, using EEG and fNIRS, the brain regions involved in three tasks using a virtual mirror therapy device (IVS4 apparatus ; Dessintey, France) implying lower limb control.

The protocol has 3 conditions :

observation (OBS), observation and imagination (OBS-IM) and observation and realization (OBS-REAL).

The order of the 3 conditions will then be randomized to avoid potential biases linked to the sequence of conditions.

The EEG recording will used the 32 channels ENOBIO apparatus. The fNIRS will used the Brite MKII apparatus

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 75 years
* Sufficient command of the French language to understand the instructions
* No known neurological medical history
* With social security coverage
* Right-handed subjects with a laterality test of Edinburgh QL> 40 (Oldfield 1971)

Exclusion Criteria:

* Minor subjects
* Adults under guardianship
* Adults under guardianship
* Pregnant or breastfeeding women
* Subjects who have objected to participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Right handed healthy subjects aged between 18 and 75 years
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Change in the EEG spectral alpha and beta-band power (8-12 and 12-30Hz) during movement (Event related Desynchronisation) | Day 0
  Beta desynchronization in dB normalized to a baseline before the movement.
Change in the beta band after movement (Beta-Rebound). | Day 0
  Beta Rebound power in dB normalized to a baseline before the movement.

SECONDARY OUTCOMES:
Mean change in the concentration of oxyhemoglobin during the task | Day 0
  Changes in the concentration of oxyhemoglobin during the task measured with Fnirs device
Mean change in the concentration of deoxyhemoglobin during the task | Day 0
  Changes in the concentration of deoxyhemoglobin during the task measured with Fnirs device

CONTACTS AND LOCATIONS:
Overall Officials: Pascal GIRAUX, Pr, Principal Investigator — CHU de Saint Etienne - Hôpital Bellevue
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Background] Bartur G, Pratt H, Frenkel-Toledo S, Soroker N. Neurophysiological effects of mirror visual feedback in stroke patients with unilateral hemispheric damage. Brain Res. 2018 Dec 1;1700:170-180. doi: 10.1016/j.brainres.2018.09.003. Epub 2018 Sep 5. PMID 30194016
- [Background] Bonnal J, Monnet F, Le BT, Pila O, Grosmaire AG, Ozsancak C, Duret C, Auzou P. Relation between Cortical Activation and Effort during Robot-Mediated Walking in Healthy People: A Functional Near-Infrared Spectroscopy Neuroimaging Study (fNIRS). Sensors (Basel). 2022 Jul 25;22(15):5542. doi: 10.3390/s22155542. PMID 35898041
- [Background] Borges LR, Fernandes AB, Melo LP, Guerra RO, Campos TF. Action observation for upper limb rehabilitation after stroke. Cochrane Database Syst Rev. 2018 Oct 31;10(10):CD011887. doi: 10.1002/14651858.CD011887.pub2. PMID 30380586
- [Background] Coll MP, Press C, Hobson H, Catmur C, Bird G. Crossmodal Classification of Mu Rhythm Activity during Action Observation and Execution Suggests Specificity to Somatosensory Features of Actions. J Neurosci. 2017 Jun 14;37(24):5936-5947. doi: 10.1523/JNEUROSCI.3393-16.2017. Epub 2017 May 30. PMID 28559380
- [Background] Fox NA, Bakermans-Kranenburg MJ, Yoo KH, Bowman LC, Cannon EN, Vanderwert RE, Ferrari PF, van IJzendoorn MH. Assessing human mirror activity with EEG mu rhythm: A meta-analysis. Psychol Bull. 2016 Mar;142(3):291-313. doi: 10.1037/bul0000031. Epub 2015 Dec 21. PMID 26689088
- [Background] Macuga KL, Frey SH. Neural representations involved in observed, imagined, and imitated actions are dissociable and hierarchically organized. Neuroimage. 2012 Feb 1;59(3):2798-807. doi: 10.1016/j.neuroimage.2011.09.083. Epub 2011 Oct 8. PMID 22005592
- [Derived] Adham A, Le BT, Bonnal J, Bessaguet H, Ojardias E, Giraux P, Auzou P. Neural basis of lower-limb visual feedback therapy: an EEG study in healthy subjects. J Neuroeng Rehabil. 2024 Jul 8;21(1):114. doi: 10.1186/s12984-024-01408-8. PMID 38978051